CLINICAL TRIAL: NCT01472393
Title: A Randomized Controlled Trial: Effects of Creatine Supplementation on Bone Mass and Turnover and Muscle Function in Healthy Postmenopausal Women
Brief Title: Creatine on Bone Mass in Postmenopausal Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Collaborators: AlzChem AG (Industry)
Responsible Party: Principal Investigator, Bruno Gualano, Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: USP.BONE
Record Dates: First submitted 2011-11-08; First posted 2011-11-16 (Estimated); Last update posted 2015-01-30 (Estimated); Status verified 2015-01

CONDITIONS: Postmenopausal Women
Keywords: creatine supplementation; bone mass; postmenopausal women; muscle function; bone markers
MeSH Terms: interventions — Creatine; Glucose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Creatine supplementation (Experimental)
  Interventions: Dietary Supplement: Creatine supplementation
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: dextrose (placebo)

INTERVENTIONS:
Dietary Supplement: Creatine supplementation — The CR group will receive either 1g or 3g of Cr monohydrate (Creapure®) per day throughout the trial. The dose of creatine will be formulated in a tablet.
  Arms: Creatine supplementation
Dietary Supplement: dextrose (placebo) — The placebo group will be given the same dose of dextrose formulated in a tablet to be consumed under the same conditions. The two types of tablets will not be distinguishable from each other having the same appearance, taste and smell.
  Arms: Placebo

SUMMARY:
Animal, in vitro and small-scale studies have suggested that creatine supplementation may augment bone mass. This clinical trial aims to investigate the effects of a 2-year creatine supplementation protocol on bone mass in postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* healthy postmenopausal women
* T-score at lumbar spine, or femoral neck or total femur of between -1SD and -2.5SD

Exclusion Criteria:

* drugs or dietary supplements that may affect bone metabolism (e.g., bisphosphonates, AINEs, hormone replacement therapy, calcium, vitamin D, creatine supplementation)
* low BMI (< 18.5 Kg/m2).

Ages: 50 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-11; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
bone mineral density (BMD) | 12 and 24 months

SECONDARY OUTCOMES:
bone markers | 12 and 24 months
  will include CTX and P1NP
history of falls | 24 months
bone microarchitecture | 12 and 24 months
muscle function | 12 and 24 months
lean mass | 12 and 24 months
laboratory parameters | 12 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Gualano, PhD, Principal Investigator — University of Sao Paulo; Rosa M Pereira, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- University of Sao Paulo - School of Medicine, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Sales LP, Pinto AJ, Rodrigues SF, Alvarenga JC, Goncalves N, Sampaio-Barros MM, Benatti FB, Gualano B, Rodrigues Pereira RM. Creatine Supplementation (3 g/d) and Bone Health in Older Women: A 2-Year, Randomized, Placebo-Controlled Trial. J Gerontol A Biol Sci Med Sci. 2020 Apr 17;75(5):931-938. doi: 10.1093/gerona/glz162. PMID 31257405
- [Derived] Lobo DM, Tritto AC, da Silva LR, de Oliveira PB, Benatti FB, Roschel H, Niess B, Gualano B, Pereira RM. Effects of long-term low-dose dietary creatine supplementation in older women. Exp Gerontol. 2015 Oct;70:97-104. doi: 10.1016/j.exger.2015.07.012. Epub 2015 Jul 17. PMID 26192975
- [Derived] Gualano B, Macedo AR, Alves CR, Roschel H, Benatti FB, Takayama L, de Sa Pinto AL, Lima FR, Pereira RM. Creatine supplementation and resistance training in vulnerable older women: a randomized double-blind placebo-controlled clinical trial. Exp Gerontol. 2014 May;53:7-15. doi: 10.1016/j.exger.2014.02.003. Epub 2014 Feb 13. PMID 24530883